CLINICAL TRIAL: NCT04228172
Title: Genotypic Influences on Network Progression in Parkinson's Disease
Status: Active, not recruiting | Type: Observational
Sponsor: Northwell Health (Other)
Collaborators: Michael J. Fox Foundation for Parkinson's Research (Other); The Silverstein Foundation for Parkinson's with GBA (Unknown)
Responsible Party: Principal Investigator, David Eidelberg, Professor & Head, Feinstein Center for Neurosciences, Feinstein Institutes for Medical Research, Northwell Health
Other Study IDs: MJFF grant 16325
Record Dates: First submitted 2020-01-07; First posted 2020-01-14 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: Parkinson's Disease
Keywords: GBA; genetic; progression; PD; glucocerebrosidase
MeSH Terms: conditions — Parkinson Disease; Disease Progression | interventions — Magnetic Resonance Spectroscopy

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Potential subjects may undergo DNA testing for GBA and LRRK2 PD mutations.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Parkinson's disease (PD) glucocerebrosidase (GBA) carriers: Parkinson's disease subjects with GBA mutation
  Interventions: Genetic: DNA/GeneticTesting; Radiation: FDG PET scan; Other: MRI scan; Other: Clinical and neuropsychological assessments
- Parkinson's disease (PD) non glucocerebrosidase (GBA) carriers: Parkinson's disease subjects without GBA mutation
  Interventions: Genetic: DNA/GeneticTesting; Radiation: FDG PET scan; Other: MRI scan; Other: Clinical and neuropsychological assessments

INTERVENTIONS:
Genetic: DNA/GeneticTesting — Subjects will be tested for GBA and LRRK2 mutation status at baseline.
Radiation: FDG PET scan — 18F-Fluoro-2-deoxy-glucose (FDG) PET scan is a nuclear medicine test that measures glucose metabolism (energy) in your brain at baseline and 18 months later.
Other: MRI scan — Magnetic Resonance Imaging (MRI) is a noninvasive scan which produces detailed pictures of the brain using a magnetic field. In addition, a special type of MRI, called resting state functional MRI (rs-fMRI), will measure and map brain activity. Conducted at baseline and 18 months later.
Other: Clinical and neuropsychological assessments — Investigator will evaluate subjects according to the Movement Disorder Society-Unified Parkinson's Disease Rating Scale (MDS-UPDRS), the standard clinical tool used to measure the severity and progression of PD. Neuropsychological evaluation will assess how one's brain functions (via pencil and paper testing), which indirectly yields information about the structural and functional integrity of the brain. Conducted at baseline and 18 months later.

SUMMARY:
In this longitudinal study, the investigators will follow Parkinson's disease (PD) patients with and without glucocerebrosidase (GBA) mutations. The investigators hypothesize that the rate of increase in brain network activity over time (network progression rate) is faster in patients with GBA gene mutations.

DETAILED DESCRIPTION:
Parkinson's disease (PD) patients with mutations in the glucocerebrosidase gene (GBA) tend to have a more aggressive disease course. GBA may therefore provide a target for disease modifying therapies in mutation carriers. Using positron emission tomography (PET) and magnetic resonance imaging (MRI) brain imaging to measure network progression rates in mutation carriers will allow for the assessment of the potential disease modifying effects of new anti-GBA therapies.

The investigators will also determine whether magnetic resonance imaging (MRI) network methods, which are less invasive and more broadly available than positron emission tomography (PET), produce comparable network progression measurements in individual patients. These determinations will be critical for the design of clinical trials of new disease-modifying drugs.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of PD made according to United Kingdom (UK) Parkinson's Disease Society Brain Bank Criteria
* Ability to provide written informed consent
* Age 40-75
* Stable dose of antiparkinsonian medication for >1 month prior to study entry

Exclusion Criteria:

* Subjects with pathogenic mutations in LRRK2 related PD mutations (subjects with variants of uncertain significance (VUS) are eligible
* History of known causative factors such as encephalitis or neuroleptic treatment
* Patients with dementia (defined as Mini-Mental Status Exam score <24 or a Telephone Interview for Cognitive Status score <26)
* Atypical parkinsonian features including oculomotor abnormalities, incontinence, ataxia, sensory loss, or pyramidal signs
* Known structural brain lesions
* Patients with history of stroke, head injury, high intracranial pressure or severe headaches
* Psychiatric disorder, including a history of major depression in the past 36 months
* Pregnant or breastfeeding women (female subjects of child-bearing potential will be screened for pregnancy before imaging).

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Study population will be recruited through local movement disorders centers in the tri-state area, prior PD studies, The Michael J. Fox Trial Finder, community outreach
Sampling Method: Non-Probability Sample
Enrollment: 32 (Estimated)
Dates: Start 2020-02-24 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-02-01 (Estimated)

PRIMARY OUTCOMES:
Increase in PD related metabolic pattern expression | Baseline and 18 months later
  Changes in PD related and PD cognition related pattern expression in 18F-2-fluoro-2-deoxy-D-glucose (FDG) PET scans
Increase in PD related functional pattern expression | Baseline and 18 months later
  Changes in PD related and PD cognition related pattern expression in resting state functional magnetic resonance imaging (rs-fMRI)

SECONDARY OUTCOMES:
Change in motor function | Baseline and 18 months later
  Change in motor function assessed with Movement Disorder Society Unified Parkinson's Disease Rating Scale (MDS-UPDRS) III (The sum score ranges between 0-132 points. Higher scores indicate more severe impairment)
Change in cognitive function | Baseline and 18 months later
  Change in cognitive function assessed with neuropsychological testing

CONTACTS AND LOCATIONS:
Overall Officials: David Eidelberg, MD, Principal Investigator — Head, Center for Neurosciences
Locations (1):
- Feinstein Institutes for Medical Research, Manhasset, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Davis MY, Johnson CO, Leverenz JB, Weintraub D, Trojanowski JQ, Chen-Plotkin A, Van Deerlin VM, Quinn JF, Chung KA, Peterson-Hiller AL, Rosenthal LS, Dawson TM, Albert MS, Goldman JG, Stebbins GT, Bernard B, Wszolek ZK, Ross OA, Dickson DW, Eidelberg D, Mattis PJ, Niethammer M, Yearout D, Hu SC, Cholerton BA, Smith M, Mata IF, Montine TJ, Edwards KL, Zabetian CP. Association of GBA Mutations and the E326K Polymorphism With Motor and Cognitive Progression in Parkinson Disease. JAMA Neurol. 2016 Oct 1;73(10):1217-1224. doi: 10.1001/jamaneurol.2016.2245. PMID 27571329
- [Background] Cilia R, Tunesi S, Marotta G, Cereda E, Siri C, Tesei S, Zecchinelli AL, Canesi M, Mariani CB, Meucci N, Sacilotto G, Zini M, Barichella M, Magnani C, Duga S, Asselta R, Solda G, Seresini A, Seia M, Pezzoli G, Goldwurm S. Survival and dementia in GBA-associated Parkinson's disease: The mutation matters. Ann Neurol. 2016 Nov;80(5):662-673. doi: 10.1002/ana.24777. Epub 2016 Oct 3. PMID 27632223
- [Background] Sidransky E, Lopez G. The link between the GBA gene and parkinsonism. Lancet Neurol. 2012 Nov;11(11):986-98. doi: 10.1016/S1474-4422(12)70190-4. PMID 23079555
- [Background] Schindlbeck KA, Eidelberg D. Network imaging biomarkers: insights and clinical applications in Parkinson's disease. Lancet Neurol. 2018 Jul;17(7):629-640. doi: 10.1016/S1474-4422(18)30169-8. PMID 29914708
- [Background] Neumann J, Bras J, Deas E, O'Sullivan SS, Parkkinen L, Lachmann RH, Li A, Holton J, Guerreiro R, Paudel R, Segarane B, Singleton A, Lees A, Hardy J, Houlden H, Revesz T, Wood NW. Glucocerebrosidase mutations in clinical and pathologically proven Parkinson's disease. Brain. 2009 Jul;132(Pt 7):1783-94. doi: 10.1093/brain/awp044. Epub 2009 Mar 13. PMID 19286695
- [Background] Winder-Rhodes SE, Evans JR, Ban M, Mason SL, Williams-Gray CH, Foltynie T, Duran R, Mencacci NE, Sawcer SJ, Barker RA. Glucocerebrosidase mutations influence the natural history of Parkinson's disease in a community-based incident cohort. Brain. 2013 Feb;136(Pt 2):392-9. doi: 10.1093/brain/aws318. PMID 23413260
- [Background] Alcalay RN, Levy OA, Waters CC, Fahn S, Ford B, Kuo SH, Mazzoni P, Pauciulo MW, Nichols WC, Gan-Or Z, Rouleau GA, Chung WK, Wolf P, Oliva P, Keutzer J, Marder K, Zhang X. Glucocerebrosidase activity in Parkinson's disease with and without GBA mutations. Brain. 2015 Sep;138(Pt 9):2648-58. doi: 10.1093/brain/awv179. Epub 2015 Jun 27. PMID 26117366
- [Background] Mazzulli JR, Xu YH, Sun Y, Knight AL, McLean PJ, Caldwell GA, Sidransky E, Grabowski GA, Krainc D. Gaucher disease glucocerebrosidase and alpha-synuclein form a bidirectional pathogenic loop in synucleinopathies. Cell. 2011 Jul 8;146(1):37-52. doi: 10.1016/j.cell.2011.06.001. Epub 2011 Jun 23. PMID 21700325
- [Background] McNeill A, Magalhaes J, Shen C, Chau KY, Hughes D, Mehta A, Foltynie T, Cooper JM, Abramov AY, Gegg M, Schapira AH. Ambroxol improves lysosomal biochemistry in glucocerebrosidase mutation-linked Parkinson disease cells. Brain. 2014 May;137(Pt 5):1481-95. doi: 10.1093/brain/awu020. Epub 2014 Feb 25. PMID 24574503
- [Background] Sardi SP, Clarke J, Viel C, Chan M, Tamsett TJ, Treleaven CM, Bu J, Sweet L, Passini MA, Dodge JC, Yu WH, Sidman RL, Cheng SH, Shihabuddin LS. Augmenting CNS glucocerebrosidase activity as a therapeutic strategy for parkinsonism and other Gaucher-related synucleinopathies. Proc Natl Acad Sci U S A. 2013 Feb 26;110(9):3537-42. doi: 10.1073/pnas.1220464110. Epub 2013 Jan 7. PMID 23297226
- [Background] Feigin A, Kaplitt MG, Tang C, Lin T, Mattis P, Dhawan V, During MJ, Eidelberg D. Modulation of metabolic brain networks after subthalamic gene therapy for Parkinson's disease. Proc Natl Acad Sci U S A. 2007 Dec 4;104(49):19559-64. doi: 10.1073/pnas.0706006104. Epub 2007 Nov 27. PMID 18042721
- [Background] Niethammer M, Eidelberg D. Metabolic brain networks in translational neurology: concepts and applications. Ann Neurol. 2012 Nov;72(5):635-47. doi: 10.1002/ana.23631. Epub 2012 Aug 31. PMID 22941893
- [Background] Eidelberg D. Metabolic brain networks in neurodegenerative disorders: a functional imaging approach. Trends Neurosci. 2009 Oct;32(10):548-57. doi: 10.1016/j.tins.2009.06.003. Epub 2009 Sep 16. PMID 19765835
- [Background] Vo A, Sako W, Fujita K, Peng S, Mattis PJ, Skidmore FM, Ma Y, Ulug AM, Eidelberg D. Parkinson's disease-related network topographies characterized with resting state functional MRI. Hum Brain Mapp. 2017 Feb;38(2):617-630. doi: 10.1002/hbm.23260. Epub 2016 May 21. PMID 27207613
- [Background] Schindlbeck, K.A. et al., Multicenter validation of disease-related Parkinson's disease pattern with resting state fMRI. 21st International Congress of Parkinson's Disease and Movement Disorders, June 8, 2018, Vancouver, Canada
- [Background] Schindlbeck, K.A. et al., Cognition-related Parkinson's disease pattern with functional MRI - Validation and clinical correlates. 62nd Congress of the German Society for Clinical Neurophysiology and Functional Imaging (DGKN), Berlin, Germany, March 15, 2018
- [Background] Huang C, Tang C, Feigin A, Lesser M, Ma Y, Pourfar M, Dhawan V, Eidelberg D. Changes in network activity with the progression of Parkinson's disease. Brain. 2007 Jul;130(Pt 7):1834-46. doi: 10.1093/brain/awm086. Epub 2007 Apr 30. PMID 17470495
- [Background] Tang CC, Poston KL, Dhawan V, Eidelberg D. Abnormalities in metabolic network activity precede the onset of motor symptoms in Parkinson's disease. J Neurosci. 2010 Jan 20;30(3):1049-56. doi: 10.1523/JNEUROSCI.4188-09.2010. PMID 20089913
- [Background] Niethammer M, Tang CC, LeWitt PA, Rezai AR, Leehey MA, Ojemann SG, Flaherty AW, Eskandar EN, Kostyk SK, Sarkar A, Siddiqui MS, Tatter SB, Schwalb JM, Poston KL, Henderson JM, Kurlan RM, Richard IH, Sapan CV, Eidelberg D, During MJ, Kaplitt MG, Feigin A. Long-term follow-up of a randomized AAV2-GAD gene therapy trial for Parkinson's disease. JCI Insight. 2017 Apr 6;2(7):e90133. doi: 10.1172/jci.insight.90133. PMID 28405611
- [Background] Spetsieris PG, Ko JH, Tang CC, Nazem A, Sako W, Peng S, Ma Y, Dhawan V, Eidelberg D. Metabolic resting-state brain networks in health and disease. Proc Natl Acad Sci U S A. 2015 Feb 24;112(8):2563-8. doi: 10.1073/pnas.1411011112. Epub 2015 Feb 9. PMID 25675473
- [Background] Mattis PJ, Tang CC, Ma Y, Dhawan V, Eidelberg D. Network correlates of the cognitive response to levodopa in Parkinson disease. Neurology. 2011 Aug 30;77(9):858-65. doi: 10.1212/WNL.0b013e31822c6224. Epub 2011 Aug 17. PMID 21849641
- [Background] Tang CC, Feigin A, Ma Y, Habeck C, Paulsen JS, Leenders KL, Teune LK, van Oostrom JC, Guttman M, Dhawan V, Eidelberg D. Metabolic network as a progression biomarker of premanifest Huntington's disease. J Clin Invest. 2013 Sep;123(9):4076-88. doi: 10.1172/JCI69411. Epub 2013 Aug 29. PMID 23985564